CLINICAL TRIAL: NCT06750796
Title: The Effect of Half Swaddling Application on Infant Sleep Routine, Maternal Sleep Quality and Postpartum Depression in Term Infants
Brief Title: The Half Swaddling Application on Infant Sleep Routine, Maternal Sleep Quality, Depression
Acronym: Half swaddling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hatice Kahyaoglu Sut, Assoc. Prof. Dr., Tanta University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Prospective controlled study
Record Dates: First submitted 2024-11-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Infant, Newborn; Maternal Outcome
Keywords: Infant; half swaddling; maternal sleep quality; postpartum depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: In this study, n=128 (64=control, 64=half swaddling group) mothers and infants who volunteered to participate in the study will be conducted in two groups as case and control, randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Other): The group that will not be treated with half swaddling
  Interventions: Behavioral: The Half Swaddling Application

INTERVENTIONS:
Behavioral: The Half Swaddling Application — Half swaddling application in term babies

SUMMARY:
In this prospective controlled study, it was aimed to examine the effects of half swaddling in term infants on infant sleep routine, maternal sleep quality and postpartum depression.

DETAILED DESCRIPTION:
In this prospective controlled study, it was aimed to examine the effects of half swaddling in term infants on infant sleep routine, maternal sleep quality and postpartum depression. half swaddling; Half swaddling applied to a newborn baby makes the baby feel completely safe as if they are still in the womb. After laying the soft fabric or baby blanket, it will be placed in the supine position. It is swaddling in a way that does not restrict the movement of the baby's arms and legs too much. n=128 (64=control, 64=half swaddling group) mothers and babies who volunteered to participate in the study will be randomized into two groups as case and control. In the half stock group; From the 1st to the 3rd month, half swaddling will be done 15 minutes before each sleep during the day. 0 (first meeting), 1, 2 and 3 months will be interviewed by phone for follow-up purposes.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old,
* Term birth (single birth over 37 weeks),
* After an uncomplicated pregnancy process, the delivery was completed by normal vaginal or cesarean delivery method,
* Not using cigarettes, alcohol and stimulants,
* BMI<30,
* Not working on night shift,
* Stable vital signs,
* Those who have not received infertility treatment,
* Do not have a chronic disease (such as hypertension, diabetes mellitus),
* Not experiencing serious depression, anxiety and stress,
* Not having any organic or non-organic disease that can cause cognitive impairment (such as Delirium, Dementia, Intellectual Retardation, etc.),
* No serious maternal complications,
* Mothers who volunteered to participate in the study will be included in the study.

For baby;

* Birth weight over 2500 g,
* Stable vital signs,
* APGAR score above 7,
* No serious neonatal complications,
* Midwives without congenital malformations will be included in the study.

Exclusion Criteria:

* under 18 years old,
* Preterm birth (under 37 weeks and/or multiple births),
* Incomplete delivery by normal vaginal or cesarean delivery method after a complicated pregnancy process,
* Using cigarettes, alcohol and stimulants,
* BMI>30,
* Working night shift,
* No stable vital signs,
* Having received infertility treatment,
* Having a chronic disease (such as hypertension, diabetes mellitus),
* Experiencing severe depression, anxiety and stress,
* Having any organic or non-organic disease that can cause cognitive impairment (such as Delirium, Dementia, Intellectual Retardation, etc.),
* Serious maternal complication,
* Mothers who do not volunteer to participate in the study will not be included in the study.

For baby;

* Birth weight of 2500 g and below,
* No stable vital signs,
* APGAR score below 7,
* Serious neonatal complication,
* Babies with congenital malformations will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum mothers
Enrollment: 128 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Follow-up telephone interview will be conducted at 0 (first interview), 1st, 2nd and 3rd months | Postpartum first 3 months
Pittsburgh Sleep Quality Index | up to 3 months
Edinburgh Postnatal Depression Scale | up to 3 months
Short Infant Sleep Routine Questionnaire | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For data privacy

REFERENCES:
- [Background] Sobaihi M, Banjari MA, Alahmadi TS. Implementation of Safe Sleep Practice Recommendations for Infants in Inpatient Wards. Cureus. 2020 Oct 25;12(10):e11155. doi: 10.7759/cureus.11155. PMID 33251063
- See also: Swaddling: Is it Safe for Your Baby? — https://www.healthychildren.org/English/ages-stages/baby/diapers-clothing/Pages/Swaddling-Is-it-Safe.aspx